CLINICAL TRIAL: NCT06222983
Title: A Prospective Cohort Study on the Efficacy and Prognosis of Surgical Intervention in Patients With Carotid Artery Stenosis
Brief Title: Efficacy and Prognosis of Surgical Intervention in Patients With Carotid Artery Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: EPSIPCS
Record Dates: First submitted 2024-01-07; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Carotid Artery Stenting; Carotid Endarterectomy; Carotid Artery Plaque
Keywords: Carotid Revascularization; Carotid Artery Stenting; Carotid Endarterectomy
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CEA group: CEA for atherosclerosis
  Interventions: Procedure: CEA or CAS
- CAS group: CEA for atherosclerosis
  Interventions: Procedure: CEA or CAS

INTERVENTIONS:
Procedure: CEA or CAS — After the patient is admitted to the hospital, the supervising doctor comprehensively evaluates the patient's general condition and adopts CEA or CAS treatment. The researcher does not provide advice to the supervising doctor and only observes safety and effectiveness

SUMMARY:
This study is a prospective, single center cohort study. By combining pathological examination of carotid atherosclerotic plaque with preoperative imaging examination, we explore the imaging characteristics of high-risk carotid plaque, and explore the effectiveness and safety of different surgical methods (CAS and CEA) for high-risk plaque patients with carotid stenosis.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 100 patients with carotid artery stenosis who underwent surgical reconstruction surgery at our research center were prospectively collected from December 2023 to December 2024. Preoperative laboratory examinations such as blood routine, biochemistry, coagulation, and imaging examinations such as carotid artery ultrasound and TCCD, carotid artery ultrasound contrast, high-resolution MRI, head MRI plain scan, carotid artery CTA or DSA were completed, Based on the comprehensive evaluation of the patient's condition by the supervising physician, the appropriate surgical method (CEA or CAS) is selected. Follow up will be conducted 1/3/6/12 months after surgery to evaluate the incidence of endpoint events (cerebral infarction+all-cause death+postoperative restenosis), MoCA and MMSE cognitive scores, quality of life scores, and severe perioperative complications. At the same time, for patients undergoing CEA surgery, pathological examination of the postoperative carotid artery plaque will be conducted to clarify the nature of the plaque, and combined with imaging examination, the characteristics of high-risk carotid artery plaques will be studied

ELIGIBILITY:
Inclusion Criteria:

1. The patient is aged 45-85 years old;
2. Symptomatic patients with stenosis degree greater than 50%, or asymptomatic patients with stenosis degree between 70% and 99% (ultrasound, CT or contrast);
3. Can complete regular follow-up;
4. The patient is informed and agrees to participate in the study.

Exclusion Criteria:

-

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with spontaneous intracranial hemorrhage within the past 12 months;
  2. Patients with larger intracranial aneurysms (diameter>5mm) that cannot be treated in advance or at the same time;
  3. Patients with chronic complete occlusion without obvious symptoms of cerebral ischemia;
  4. Patients with severe dementia;
  5. Carotid artery opening lesion;
  6. Severe intracranial serial stenosis lesions;
  7. Carotid artery dissection;
  8. Lesions with combined carotid artery aneurysm;
  9. Patients with generally poor physical condition who cannot tolerate surgery;
  10. Coagulation dysfunction, contraindications to heparin and antiplatelet drugs;
  11. Patients who are participating in clinical trials of other drugs or devices but have not reached the trial endpoint;
  12. Pregnant and lactating women;
  13. The researchers believe that patients who are not suitable to participate in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Any Periprocedural Stroke, Myocardial Infarction, or Death During1 month Peri-procedural Period, and Postprocedural Ipsilateral Stroke 1 to 12-months. | 0 to 12 months
  Composite of any periprocedural stroke (ipsilateral or contralateral; major or minor), myocardial infarction, or death during1 month peri-procedural period, and postprocedural ipsilateral stroke 1 to 12-months.
Rate of complications | 30days
  Rate of complications within 30 days, complications include cranial nerve and peripheral nerve injury, vascular injury, wound complications as neck incision or related to puncture site, and other (such as anesthesia) complications.
Incidence of ipsilateral stroke | 30days
  Incidence of ipsilateral stroke at 30 days follow up
Incidence of death | 30 days
  Incidence of death at 30 days follow up.
Carotid restenosis rate | 3,6,12 months
  Carotid restenosis was defined as restenosis ≥50% after carotid revascularization, that is, peak systolic velocity ratio (PSVR) ≥2.0 on ultrasound examination.
Improvement in cognitive function | 0,3,6,12months
  Cognitive function was assessed by Mini-mental State Examination (MMSE) during follow up.
Improvement in cognitive function | 0,3,6,12months
  Cognitive function was assessed by Montreal Cognitive Assessment Scale (MoCA) during follow up.
Quality of life rating | 30 days
  Use VascuQol to evaluate quality of life scores

SECONDARY OUTCOMES:
Ultrasound and pathological indicators related to high-risk plaques | 0-7days
  Ultrasound are used to visualize plaques, combined with pathological examination, to identify the imaging characteristics of high-risk plaques
CT and pathological indicators related to high-risk plaques | 0-7days
  CT are used to visualize plaques, combined with pathological examination, to identify the imaging characteristics of high-risk plaques
MRI and pathological indicators related to high-risk plaques | 0-7days
  MRI are used to visualize plaques, combined with pathological examination, to identify the imaging characteristics of high-risk plaques

CONTACTS AND LOCATIONS:
Overall Officials: Lianrui Guo, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided